CLINICAL TRIAL: NCT00641615
Title: Phase I Study of Peptide Vaccine and S-1 Plus CPT-11 Chemotherapy in Patients With Unresectable Recurrent or Metastatic Colorectal Cancer
Brief Title: Peptide Vaccine and S-1/CPT-11 Therapy for Patients With Unresectable Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kazuhiko Yoshimatsu (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Sponsor-Investigator, Kazuhiko Yoshimatsu, Ascociate professor of surgery, Tokyo Women's Medical University
Organization: Tokyo Women's Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWMU1035
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1 (Experimental)
  Interventions: Biological: RNF43-721

INTERVENTIONS:
Biological: RNF43-721 — Doses of 0.5mg, 1.0mg, 3.0mg/body/week
  Other Names: S-1/CPT-11

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of different doses of RNF43-721 emulsified with Montanide ISA 51 in combination with S-1/CPT-11 chemotherapy.

DETAILED DESCRIPTION:
RNF43 is a cancer testis antigen which express widely in colorectal cancer tissue but not in normal organs. RNF43-721 induces HLA A24 restricted specific cytotoxic T lymphocytes (CTL) against RNF43 expressed target. S-1/CPT-11 chemotherapy is performed unresectable advanced colorectal cancer in Japan and is reported to be obtained almost the same result compared with FOLFOX or FOLFIRI as first-line chemotherapy for advanced colorectal cancer. Because synergistic effect between vaccine therapy and chemotherapy will be expected, we plan phase I study to evaluate the safety and immune response of different doses of RNF43-721 emulsified with Montanide ISA 51 in combination with S-1/CPT-11 chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-1
* Life expectancy > 3 months
* HLA A24 positive
* Histologically diagnosed as colorectal cancer with measurable lesion
* Laboratory values as follows:WBC>3000/mm3, Hb>10mg/dl, Plt>75000/mm3, Creatinine<1.2mg/dl, T. bil.<1.5mg/dl, AST, ALT<3x normal limits
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Active other malignancy
* Active infection
* Immune deficiency
* Current treatment with steroids and immunosuppressive agents
* Pregnancy and breast feeding
* Inability oral intake
* Psychic disease
* Hepatitis B, C virus
* HIV infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety (toxicities as assessed by NCI CTCAE version 3) | 2 months

SECONDARY OUTCOMES:
Specific CTL induction in vitro, Objective rate as assessed by RECST criteria | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiko Yoshimatsu, MD, Principal Investigator — Tokyo Women's Medical University Medical Center East
Locations (1):
- Tokyo Women's Medical University Medical Center East, Tokyo, Japan

REFERENCES:
- [Background] Uchida N, Tsunoda T, Wada S, Furukawa Y, Nakamura Y, Tahara H. Ring finger protein 43 as a new target for cancer immunotherapy. Clin Cancer Res. 2004 Dec 15;10(24):8577-86. doi: 10.1158/1078-0432.CCR-04-0104. PMID 15623641
- [Background] Yoshimatsu K, Yokomizo H, Fujimoto T, Umehara A, Otani T, Matsumoto A, Osawa G, Ogawa K. Pilot study of simplified low-dose S-1 plus CPT-11 as first-line chemotherapy for patients with advanced colorectal cancer. Anticancer Res. 2007 May-Jun;27(3B):1657-61. PMID 17595792